CLINICAL TRIAL: NCT03189563
Title: A Phase IIa, Randomized, Multicenter, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Efficacy of DA-9805 in Subjects With Parkinson's Disease
Brief Title: Safety and Efficacy of DA-9805 for Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA-9805-PD-001
Record Dates: First submitted 2017-06-12; First posted 2017-06-16 (Actual); Results first posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — DA-9805

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): placebo, tid
  Interventions: Other: Placebo
- DA-9805 low (Experimental): DA-9805 45mg
  Interventions: Drug: DA-9805 45mg
- DA-9805 high (Experimental): DA-9805 90mg
  Interventions: Drug: DA-9805 90mg

INTERVENTIONS:
Drug: DA-9805 45mg — DA-9805 15mg tid
  Other Names: DA-9805
  Arms: DA-9805 low
Drug: DA-9805 90mg — DA-9805 30mg tid
  Other Names: DA-9805
  Arms: DA-9805 high
Other: Placebo — Placebo, tid
  Arms: Placebo

SUMMARY:
This is a phase IIa, first in human, randomized, double-blind, multicenter study to evaluate the safety, tolerability and efficacy of DA-9805 at 45mg, 90mg versus placebo in subjects diagnosed with early Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is recognized as one of the most common neurologic disorders, affecting approximately 1% of individuals older than 60 years. There are 2 major neuropathologic findings: the loss of pigmented dopaminergic neurons in the substantia nigra pars compacta (SNpc) and the presence of Lewy bodies.

Parkinson's disease affects an estimated 1.5 million persons in the United States, with over ten million affected worldwide, and these estimates are expected to increase substantially in the next few decades. Despite the increasing prevalence, the approved agents for the early management of Parkinson's disease have changed little in the past decade; however, there have been advances in drug delivery, dosing, and the use of combination therapy in an attempt to reduce adverse events. The most important, unmet medical need in targeting Parkinson's disease is developing agents with neuroprotective potential. So far, no drug has been shown to reduce or slow down the progression of PD.

DA-9805 is a botanical drug product composed of three main raw herbal materials. It is expected that DA-9805 will help treat PD by prevention of dopaminergic neurodegeneration via recovery of mitochondrial dysfunction, anti-inflammatory effect and relief from Endoplasmic reticulum (ER) stress and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are between 30 and 79 years old inclusive with a clinical diagnosis of Parkinson's disease as per UK Brain Bank Criteria for two (2) years or less at screening.
* Hoehn and Yahr I or II at screening.
* Subjects who are newly diagnosed & currently not on any Parkinson's disease medication (or) subjects who are on stable doses for at least 4 weeks prior to screening on Amantadine or anticholinergics for treatment of Parkinson's disease

  *Note: Subjects that had anti-parkinsonian medication (including levodopa, dopamine agonists, entacapone and monoamine oxidase-B inhibitors) discontinued at least 60 days prior to screening, e.g., for intolerance, may be considered eligible if all other eligibility requirements are met.
* Women of child-bearing potential should use reliable contraception. Acceptable methods of contraception include: surgical sterilization (e.g. bilateral tubal ligation), hormonal contraception (implantable, patch, and oral), and double-barrier methods (condom, diaphragm and spermicide are each considered a barrier). Women of child-bearing potential are defined as women physiologically capable of becoming pregnant, UNLESS they meet the following criteria:

  (1)Post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum Follicle Stimulating Hormone (FSH) levels > 40mIU/m, OR; (2)6 weeks post surgical bilateral oophorectomy with or without hysterectomy
* If a male and heterosexually active with a female of childbearing potential, the subject must agree to use a double barrier method of birth control (or must have been surgically sterilized) and to not donate sperm during the study.
* Without clinically significant abnormalities in physical exam, neurological exam and laboratory assessments (urine/blood routine, biochemical tests and ECG) which would exclude the subject from the study in the opinion of the Investigator. For Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) the screening levels should be ≤ 2 times upper limit normal
* Subject is capable of providing informed consent and is willing to sign the ICF prior to study Screening and agrees to comply with the study protocol requirements.

Exclusion Criteria:

* Subject has an atypical parkinsonian syndrome or secondary parkinsonism (e.g., due to drugs, metabolic neurogenetic disorders, encephalitis, cerebrovascular disease or degenerative disease).
* Subjects with history of neurosurgical intervention for Parkinson's disease.
* Subjects who meet the DSM-V criteria at screening for bipolar disorder, major depressive disorder, psychotic disorders, or any other comorbid mental disorders that in the opinion of the Investigator may interfere with study conduct and results interpretation.
* Subjects with clinical diagnosis of dementia (MMSE score <24) as determined by the investigator using Mini-Mental State Examination (MMSE).
* Female subjects who are pregnant or breast feeding.
* Initiation of any anti-parkinsonian medication (including levodopa, dopamine agonists, entacapone and monoamine oxidase-B inhibitors) for the duration of the trial.
* Initiation of Amantadine or anticholinergics for newly diagnosed subjects or change in the dosage of Amantadine or anticholinergics during the trial for subjects who were on stable doses for 4 weeks prior to screening.
* Subjects who used investigational drugs or devices within 60 days prior to screening or investigational biologics within the last 6 months prior to screening.
* Subjects with a clinically significant or surgical condition, including major surgeries within 28 days prior to enrollment

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sotirios A Parashos, MD, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Institute, Bloomington, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | DA-9805 Low | DA-9805 High
Started | 20 | 21 | 20
ITT Population | 20 | 21 | 19
Safety Population | 20 | 21 | 19
Completed | 19 | 20 | 18
Not Completed | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | DA-9805 Low | DA-9805 High | Total
Number analyzed (Participants) | 20 | 21 | 19 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (7.30) | 61.9 (9.24) | 64.2 (9.36) | 64.2 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 9 | 23
  Male | 13 | 14 | 10 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 17 | 19 | 19 | 55
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (6.12) | 28.1 (6.61) | 27.1 (4.23) | 27.9 (5.72)

OUTCOME MEASURES:

1. Primary Outcome: Change in Motor MDS-UPDRS Score From Baseline at Week 12
Description: Analysis of the Change from Baseline in the sum of the Movement Disorders Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) Part II, Part III and Part IV at week 12. (Change from baseline = Post Baseline Measurement - Baseline Measurement) MDS-UPDRS is a multimodal scale assessing both impairment and disability and is separated into 4 subscales.
  Each parkinsonian sign or symptom is rated on a 5-point severity scale (ranging from 0 to 4).
  The maximum total UPDRS score is 272, indicating the worst possible disability from PD.
  Part I: This assesses non-motor experiences of daily living (13 items, Score range: 0~52) Part II: This assesses motor experiences of daily living (13 items, Score range: 0~52) Part III: This assesses the motor signs of PD (33 items, Score range: 0~132) Part IV: This assesses motor complications, dyskinesias and motor fluctuations using historical and objective information (6 items, Score range: 0~26)
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | DA-9805 Low | DA-9805 High
Number analyzed (Participants) | 20 | 21 | 19
score on a scale | 1.4 (5.56) | -0.9 (7.03) | -1.2 (8.41)
Statistical Analysis 1: Comparison: Placebo vs DA-9805 Low; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.3656, ANCOVA — p-value is from ANCOVA model adjusted for baseline motor MDS-UPDRS total score. All statistical tests for efficacy are two-sided tests, with α=0.05
Statistical Analysis 2: Comparison: Placebo vs DA-9805 High; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.3119, ANCOVA — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change in Total MDS- UPDRS Score
Description: Analysis of the Change from Baseline in the sum of the Movement Disorders Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) Part I, Part II, Part III and Part IV at week 12. (Change from baseline = Post Baseline Measurement - Baseline Measurement) MDS-UPDRS is a multimodal scale assessing both impairment and disability and is separated into 4 subscales.
  Each parkinsonian sign or symptom is rated on a 5-point severity scale (ranging from 0 to 4).
  The maximum total UPDRS score is 272, indicating the worst possible disability from PD.
  Part I: This assesses non-motor experiences of daily living (13 items, Score range: 0~52) Part II: This assesses motor experiences of daily living (13 items, Score range: 0~52) Part III: This assesses the motor signs of PD (33 items, Score range: 0~132) Part IV: This assesses motor complications, dyskinesias and motor fluctuations using historical and objective information (6 items, Score range: 0~26)
Time Frame: 12 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Placebo | DA-9805 Low | DA-9805 High
Number analyzed (Participants) | 20 | 21 | 19
score | 1.6 (7.15) | -2.4 (7.91) | -1.7 (9.16)
Statistical Analysis 1: Comparison: Placebo vs DA-9805 Low; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.1470, ANCOVA — p-value is from ANCOVA model adjusted for baseline MDS-UPDRS total score. All statistical tests for efficacy are two-sided tests, with α=0.05
Statistical Analysis 2: Comparison: Placebo vs DA-9805 High; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.2520, ANCOVA — [p-value comment as in outcome 2, analysis 1]

3. Secondary Outcome: Change in MDS-UPDRS Subscale scores_Part I
Description: Analysis of the Change from Baseline in the sum of the Movement Disorders Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) Part I at week 12. (Change from baseline = Post Baseline Measurement - Baseline Measurement) MDS-UPDRS is a multimodal scale assessing both impairment and disability and is separated into 4 subscales.
  Each parkinsonian sign or symptom is rated on a 5-point severity scale (ranging from 0 to 4).
  The maximum total UPDRS score is 272, indicating the worst possible disability from PD.
  Part I: This assesses non-motor experiences of daily living (13 items, Score range: 0~52) Part II: This assesses motor experiences of daily living (13 items, Score range: 0~52) Part III: This assesses the motor signs of PD (33 items, Score range: 0~132) Part IV: This assesses motor complications, dyskinesias and motor fluctuations using historical and objective information (6 items, Score range: 0~26)
Time Frame: 12 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | DA-9805 Low | DA-9805 High
Number analyzed (Participants) | 20 | 21 | 19
score on a scale | 0.1 (3.3) | -1.3 (2.82) | -0.5 (3.04)
Statistical Analysis 1: Comparison: Placebo vs DA-9805 Low; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.1528, ANCOVA — p-value is from ANCOVA model adjusted for baseline MDS-UPDRS part 1 subscale score. All statistical tests for efficacy are two-sided tests, with α=0.05
Statistical Analysis 2: Comparison: Placebo vs DA-9805 High; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.6146, ANCOVA — [p-value comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change in S&E Total Score
Description: Change in Schwab and England (S&E) Scale total score from baseline at week 12. (Change from baseline = Post Baseline Measurement - Baseline Measurement) The Schwab & England Activities of Daily Living (ADL) scale reflects the speed, ease, and independence with which an individual performs daily activities, or personal chores, such as eating, toileting, and dressing. This scale uses a rating scale from 0% to 100%, with 100% representing complete independence in performing daily activities and 0% representing a vegetative, bedridden state.
Time Frame: 12 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | DA-9805 Low | DA-9805 High
Number analyzed (Participants) | 20 | 21 | 19
score on a scale | 2.0 (8.34) | 1.0 (7.00) | 0.5 (5.24)
Statistical Analysis 1: Comparison: Placebo vs DA-9805 Low; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.5691, ANCOVA — p-value is from ANCOVA model adjusted for baseline S&E scale total score. All statistical tests for efficacy are two-sided tests, with α=0.05
Statistical Analysis 2: Comparison: Placebo vs DA-9805 High; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.1309, ANCOVA — [p-value comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change in PDQ-39 Score- Summary Index
Description: Change in Parkinson's Disease Questionnaire (PDQ-39) total score from baseline at week 12.(Change from baseline = Post Baseline Measurement - Baseline Measurement) The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing eight domains of health (mobility [10 items], activities of daily living [6 items], emotional wellbeing [6 items], stigma [4 items], cognition [4 items], social support [3 items], communication [3 items] and bodily discomfort [3 items]) which subjects consider to be adversely affected by the disease.
  Each item is scored on the following 5-point scale. The PDQ-39 Summary Index (PDQ-SI) is the sum of all answers divided by the highest score possible (i.e., number of answers multiplied by 4) which is multiplied by 100 to put the score on a 0 - 100 scale where lower scores indicate a better perceived health status and higher scores are ass
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | DA-9805 Low | DA-9805 High
Number analyzed (Participants) | 20 | 21 | 19
score on a scale | -1.3 (4.95) | -1.7 (4.58) | -1.5 (4.57)
Statistical Analysis 1: Comparison: Placebo vs DA-9805 Low; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.7913, ANCOVA — p-value is from ANCOVA model adjusted for baseline PDQ-39 summary index. All statistical tests for efficacy are two-sided tests, with α=0.05
Statistical Analysis 2: Comparison: Placebo vs DA-9805 High; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.9399, ANCOVA — [p-value comment as in outcome 5, analysis 1]

6. Secondary Outcome: Change in H&Y Total Score at Week 12
Description: Change in Hoehn and Yahr (H&Y) scale total score from baseline at week 12. (Change from baseline = Post Baseline Measurement - Baseline Measurement) H&Y describes five stages to PD progression (Score 1~5). A lower score represent a lower amount of symptoms.
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | DA-9805 Low | DA-9805 High
Number analyzed (Participants) | 20 | 21 | 19
score on a scale | 0.1 (0.39) | 0.0 (0.59) | 0.1 (0.46)
Statistical Analysis 1: Comparison: Placebo vs DA-9805 Low; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.4978, ANCOVA — p-value is from ANCOVA model adjusted for baseline H&Y scale total score. All statistical tests for efficacy are two-sided tests, with α=0.05
Statistical Analysis 2: Comparison: Placebo vs DA-9805 High; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.8880, ANCOVA — [p-value comment as in outcome 6, analysis 1]

7. Secondary Outcome: Change in MDS-UPDRS Subscale scores_Part II
Description: Analysis of the Change from Baseline in the sum of the Movement Disorders Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) Part II at week 12. (Change from baseline = Post Baseline Measurement - Baseline Measurement) MDS-UPDRS is a multimodal scale assessing both impairment and disability and is separated into 4 subscales.
  Each parkinsonian sign or symptom is rated on a 5-point severity scale (ranging from 0 to 4).
  The maximum total UPDRS score is 272, indicating the worst possible disability from PD.
  Part I: This assesses non-motor experiences of daily living (13 items, Score range: 0~52) Part II: This assesses motor experiences of daily living (13 items, Score range: 0~52) Part III: This assesses the motor signs of PD (33 items, Score range: 0~132) Part IV: This assesses motor complications, dyskinesias and motor fluctuations using historical and objective information (6 items, Score range: 0~26)
Time Frame: 12 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | DA-9805 Low | DA-9805 High
Number analyzed (Participants) | 20 | 21 | 19
score on a scale | 0.8 (3.05) | 1.3 (2.26) | -0.6 (3.67)
Statistical Analysis 1: Comparison: Placebo vs DA-9805 Low; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.5755, ANCOVA — p-value is from ANCOVA model adjusted for baseline MDS-UPDRS part 2 subscale score. All statistical tests for efficacy are two-sided tests, with α=0.05
Statistical Analysis 2: Comparison: Placebo vs DA-9805 High; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.1517, ANCOVA — [p-value comment as in outcome 7, analysis 1]

8. Secondary Outcome: Change in MDS-UPDRS Subscale scores_Part III
Description: Analysis of the Change from Baseline in the sum of the Movement Disorders Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) Part III at week 12. (Change from baseline = Post Baseline Measurement - Baseline Measurement) MDS-UPDRS is a multimodal scale assessing both impairment and disability and is separated into 4 subscales.
  Each parkinsonian sign or symptom is rated on a 5-point severity scale (ranging from 0 to 4).
  The maximum total UPDRS score is 272, indicating the worst possible disability from PD.
  Part I: This assesses non-motor experiences of daily living (13 items, Score range: 0~52) Part II: This assesses motor experiences of daily living (13 items, Score range: 0~52) Part III: This assesses the motor signs of PD (33 items, Score range: 0~132) Part IV: This assesses motor complications, dyskinesias and motor fluctuations using historical and objective information (6 items, Score range: 0~26)
Time Frame: 12 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | DA-9805 Low | DA-9805 High
Number analyzed (Participants) | 20 | 21 | 19
score on a scale | 0.7 (5.0) | -1.7 (6.21) | -0.6 (6.02)
Statistical Analysis 1: Comparison: Placebo vs DA-9805 Low; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.2095, ANCOVA — p-value is from ANCOVA model adjusted for baseline MDS-UPDRS part 3 subscale score. All statistical tests for efficacy are two-sided tests, with α=0.05
Statistical Analysis 2: Comparison: Placebo vs DA-9805 High; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.6094, ANCOVA — [p-value comment as in outcome 8, analysis 1]

9. Secondary Outcome: Change in MDS-UPDRS Subscale scores_Part IV
Description: Analysis of the Change from Baseline in the sum of the Movement Disorders Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) Part IV at week 12. (Change from baseline = Post Baseline Measurement - Baseline Measurement) MDS-UPDRS is a multimodal scale assessing both impairment and disability and is separated into 4 subscales.
  Each parkinsonian sign or symptom is rated on a 5-point severity scale (ranging from 0 to 4).
  The maximum total UPDRS score is 272, indicating the worst possible disability from PD.
  Part I: This assesses non-motor experiences of daily living (13 items, Score range: 0~52) Part II: This assesses motor experiences of daily living (13 items, Score range: 0~52) Part III: This assesses the motor signs of PD (33 items, Score range: 0~132) Part IV: This assesses motor complications, dyskinesias and motor fluctuations using historical and objective information (6 items, Score range: 0~26)
Time Frame: 12 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | DA-9805 Low | DA-9805 High
Number analyzed (Participants) | 20 | 21 | 19
score on a scale | 0.3 (1.38) | -0.1 (0.45) | 0.0 (0.00)
Statistical Analysis 1: Comparison: Placebo vs DA-9805 Low; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.2260, ANCOVA — p-value is from ANCOVA model adjusted for baseline MDS-UPDRS part 4 subscale score. All statistical tests for efficacy are two-sided tests, with α=0.05
Statistical Analysis 2: Comparison: Placebo vs DA-9805 High; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.2260, ANCOVA — p-value is from ANCOVA model adjusted for baseline MDS-UPDRS part 4 subscale score All statistical tests for efficacy are two-sided tests, with α=0.05

10. Secondary Outcome: Change in Clinical Global Impression-Severity (CGI-S)
Description: The Global Impression-Severity (CGI) measures global severity of illness at a given point in time, and the improvement from baseline at visits following the initial baseline visit. (Change from baseline = Post Baseline Measurement - Baseline Measurement) At the screening and baseline visit, the investigator assessed the severity on a seven-point scale. At subsequent visits, the investigator was to assess the subject's severity (CGI-S) and improvement (CGI-I) relative to baseline.
  Severity of Illness (CGI-S) Rating should account for severity of the patient's illness. 0 = Not assessed
  1. = Normal, not at all ill
  2. = Borderline ill
  3. = Mildly ill
  4. = Moderately ill
  5. = Markedly ill
  6. = Severely ill
  7. = Extremely ill
Time Frame: 12 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | DA-9805 Low | DA-9805 High
Number analyzed (Participants) | 20 | 21 | 19
score on a scale | 0.1 (0.60) | 0.0 (0.67) | 0.1 (0.71)
Statistical Analysis 1: Comparison: Placebo vs DA-9805 Low; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.8274, ANCOVA — p-value is from ANCOVA model adjusted for baseline CGI-S score. All statistical tests for efficacy are two-sided tests, with α=0.05
Statistical Analysis 2: Comparison: Placebo vs DA-9805 High; Change from baseline is based on subjects with paired values; Test type: Superiority; p = 0.3416, ANCOVA — [p-value comment as in outcome 10, analysis 1]

11. Secondary Outcome: Scores of Clinical Global Impression-Improvement (CGI-I)
Description: The Global Impression-Severity (CGI) measures global severity of illness at a given point in time, and the improvement from baseline at visits following the initial baseline visit.
  At the screening and baseline visit, the investigator assessed the severity on a seven-point scale. At subsequent visits, the investigator was to assess the subject's severity (CGI-S) and improvement (CGI-I) relative to baseline.
  Global Improvement (CGI-I):
  Compared to the patient's condition at the baseline of this study, how much has the patient's illness improved or worsened? 0 = Not assessed
  1. = Very much improved
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse
Time Frame: 12 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | DA-9805 Low | DA-9805 High
Number analyzed (Participants) | 20 | 21 | 19
score on a scale | 3.6 (0.69) | 3.8 (0.54) | 3.9 (1.12)
Statistical Analysis 1: Comparison: Placebo vs DA-9805 Low; Test type: Superiority; p = 0.4052, ANCOVA — P-value is from ANCOVA model. All statistical tests for efficacy are two-sided tests, with α=0.05
Statistical Analysis 2: Comparison: Placebo vs DA-9805 High; Test type: Superiority; p = 0.2643, ANCOVA — P-value is from ANCOVA model. All statistical tests for efficacy are two-sided tests, with α=0.05

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Placebo | DA-9805 Low | DA-9805 High
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 2/21 | 0/19
Other Adverse Events (participants affected / at risk) | 11/20 | 8/21 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | DA-9805 Low (N=21) | DA-9805 High (N=19)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
STRESS CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | DA-9805 Low (N=21) | DA-9805 High (N=19)
tremor (Nervous system disorders) | 1 (1) | 1 (1) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (2)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT03189563/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT03189563/SAP_001.pdf